CLINICAL TRIAL: NCT06531993
Title: Effect of Pectin in Chronic Kidney Disease Patients ( Stage 3 and 4 )
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maha Gamal Mahmoud Ahmed, Resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pectin in CKD
Record Dates: First submitted 2024-06-10; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Pectins

STUDY DESIGN:
Intervention Model Description: Pectin, a class of heteropolysaccharides based on polygalacturonic acid, is a safe and non-toxic natural food additive recommended by the Joint FAO/WHO Committee on Food Additives with no daily additive limit . Pectin is mainly obtained from apple pomace, citrus peels and sugar beets, ancurrently, commercial pectin contains ≥65% Gal-A (galacturonic acid)
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pectin group (Active Comparator): Pectin treatment
  Interventions: Drug: Pectin
- Placepo group (Placebo Comparator): Standard of care
  Interventions: Drug: Pectin

INTERVENTIONS:
Drug: Pectin — Using pectin as tablets 600 mg per day for 6 months

SUMMARY:
Effect of pectin in chronic kidney disease patients

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a serious global health problem leading to serious comorbidities, end-stage renal disease (ESRD), and death

From 1990 to 2016, the prevalence of CKD increased by 90% worldwide, which is closely tied to the increase in at-risk populations with diabetes mellitus (DM), hypertension (HTN), and prediabetes . It is estimated to be around 9.1 to 13.4%. This means there are about 700 million to over 800 million cases of CKD worldwide.

In 2017, CKD resulted in 1.2 million deaths and was the 12th leading cause of death worldwide . And in the same year, the estimated prevalence of CKD in Egypt was 7.1 million individuals, which means 106 patients/1000 population .

Pectin, a class of heteropolysaccharides based on polygalacturonic acid, is a safe and non-toxic natural food additive recommended by the Joint FAO/WHO Committee on Food Additives with no daily additive limit . Pectin is mainly obtained from apple pomace, citrus peels and sugar beets, ancurrently, commercial pectin contains ≥65% Gal-A (galacturonic acid).

Among the patients who tried to take the pectin, unexpectedly was found that the pectin had a significant effect on the rapid reduction of blood creatinine concentration in patients with chronic kidney disease. So, the authors followed up the physical examination indeces of chronic kidney disease patients who took the Pectin .

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of CKD patients (stage 3 and 4)
2. age between 18 and 60 years
3. Must be able to swallow tablets

Exclusion Criteria:

1- End stage renal disease ( stage 5 ) 2 - Patients with renal transplantation 3- pregnancy 4- Presence of malignancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 98 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
effect of pectin in GFR improvement in ckd patients | 6 month
  Measure eGFR using CKD epi equation,

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Anwer Thabet, Study Director — Prof

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.efsa.europa.eu/en/efsajournal/pub/4866
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6341125/
- See also: Related Info — http://dx.doi.org/10.21203/rs.3.rs-3689543/v1